CLINICAL TRIAL: NCT06899672
Title: Analyzing the Effect of Disinfection Additives on the Linear Dimensional Stability of Dental Alginate Impressions: A Quasi-Experimental Comparative Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Dr. Aiman yaseen, Bachelor of Dental Surgery, Altamash Institute of Dental Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AIDM/ERC/10/2024/01
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Dimensional Changes
MeSH Terms: interventions — Chlorhexidine; Alginates; Chitosan; Silver Nitrate; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Control Group (Distilled Water) (Experimental): Participants (specimens) will receive alginate mixed with distilled water without any disinfectant, serving as the baseline group
  Interventions: Other: Alginate mixed with distilled water
- CHX Group (0.2% Chlorhexidine) (Experimental): Participants (specimens) will receive alginate mixed with 0.2% Chlorhexidine solution to assess its effect on dimensional stability
  Interventions: Other: 0.2% Chlorhexidine + Alginate
- Chitosan Group (1% Chitosan) (Experimental): Participants (specimens) will receive alginate mixed with 1% Chitosan solution to evaluate its effect on dimensional stability
  Interventions: Other: 1% Chitosan + Alginate
- Silver Nitrate Group (0.2% Silver Nitrate) (Experimental): Participants (specimens) will receive alginate mixed with 0.2% Silver Nitrate solution to evaluate its effect on dimensional stability
  Interventions: Other: 0.2% Silver Nitrate + Alginate
- Silver Nanoparticles Group (Green-Synthesized AgNPs) (Experimental): Participants (specimens) will receive alginate mixed with green-synthesized silver nanoparticles to investigate its impact on dimensional stability
  Interventions: Other: Green-synthesized Silver Nanoparticles + Alginate
- PVP-Iodine Group (15% Povidone-Iodine) (Experimental): Participants (specimens) will receive alginate mixed with 15% Povidone-Iodine solution to determine its effect on dimensional stability
  Interventions: Other: 15% Povidone-Iodine + Alginate

INTERVENTIONS:
Other: Alginate mixed with distilled water — Alginate will be mixed with distilled water only, without any disinfectant additive, to serve as the control for comparison
  Arms: Control Group (Distilled Water)
Other: 0.2% Chlorhexidine + Alginate — Alginate will be mixed with 0.2% Chlorhexidine solution to evaluate its effect on the linear dimensional stability of alginate impressions
  Arms: CHX Group (0.2% Chlorhexidine)
Other: 1% Chitosan + Alginate — Alginate will be mixed with 1% Chitosan solution to assess its influence on the linear dimensional stability of alginate impressions
  Arms: Chitosan Group (1% Chitosan)
Other: 0.2% Silver Nitrate + Alginate — Alginate will be mixed with 0.2% Silver Nitrate solution to determine its effect on the dimensional stability of alginate impressions
  Arms: Silver Nitrate Group (0.2% Silver Nitrate)
Other: Green-synthesized Silver Nanoparticles + Alginate — Alginate will be mixed with a solution of green-synthesized Silver Nanoparticles to investigate its effect on the dimensional stability of alginate impressions
  Arms: Silver Nanoparticles Group (Green-Synthesized AgNPs)
Other: 15% Povidone-Iodine + Alginate — Alginate will be mixed with 15% Povidone-Iodine solution to analyze its influence on the dimensional stability of alginate impressions
  Arms: PVP-Iodine Group (15% Povidone-Iodine)

SUMMARY:
This quasi-experimental comparative study investigates the effects of incorporating various self-disinfecting agents-0.2% Chlorhexidine (CHX), 1% Chitosan solution, 0.2% Silver Nitrate (AgNO3), green-synthesized Silver Nanoparticles (AgNPs), and 15% PVP-Iodine-on the linear dimensional stability of dental alginate impressions. Alginate is widely used in dentistry but is prone to dimensional changes and contamination. This study aims to assess whether integrating these disinfectants can reduce microbial risks without compromising the material's dimensional accuracy, thereby improving infection control and the precision of dental prostheses

ELIGIBILITY:
Inclusion Criteria:

* Dental stone casts free from excessive porosity, fractures, or other visible defects that could affect dimensional stability measurements.
* Typodont models with intact maxillary arch configurations.

Exclusion Criteria:

* Distorted impressions, under-extended impressions, impressions that detach from the tray before pouring, and impressions with voids, on visual inspection.
* Dental cast with a fracture component, incomplete pouring, and those with voids or bubbles.

Min Age: 60 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Linear Dimensional Stability of Alginate Impressions | 1 hour after impression making and cast pouring
  Measurement of the linear dimensional changes (in millimeters) of alginate impressions mixed with disinfectant additives compared to the control group.